CLINICAL TRIAL: NCT02020018
Title: Negative Pressure Wound Therapy for Prevention of Wound Infection After Heart Surgery
Brief Title: Negative Pressure Wound Therapy for Prevention of Poststernotomy Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Principal Investigator, Hartzell V. Schaff, Professor of Surgery, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-007901
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective group (Experimental): Negative pressure wound therapy (Prevena Incision Management System) applied immediately postoperatively.
  Interventions: Device: Prevena Incision Management System
- Retrospective arm (Active Comparator): Conventional sterile dry wound dressing applied immediately postoperatively.
  Interventions: Other: Conventional sterile dry wound dressing

INTERVENTIONS:
Device: Prevena Incision Management System — negative pressure therapy that will be applied instead of the regular dressing immediately postoperatively in high risk patients and kept for 6-7 days
  Other Names: negative pressure therapy; wound VAC; Prevena
  Arms: Prospective group
Other: Conventional sterile dry wound dressing — regular dressing that is applied immediately postoperatively for high risk patients in the operating room after sternotomy
  Other Names: poststernotomy wound dressing; standard dressing after sternotomy
  Arms: Retrospective arm

SUMMARY:
This prospective study evaluates the role of negative pressure wound therapy or wound VAC as a dressing over the incision to prevent poststernotomy wound infection in high risk patients.

DETAILED DESCRIPTION:
Surgical site infection after cardiac surgery is a major cause for increased morbidity and mortality. Vacuum assisted closure (VAC) has been used in the management of open and infected wounds. However, its effectiveness as a prophylactic measure for prevention of surgical site infection after routine cardiac surgery is unknown.

ELIGIBILITY:
Inclusion criteria:

1. Transplant patients
2. BMI >30
3. Type I (insulin-dependent) diabetics
4. Severe chronic obstructive pulmonary disease (COPD)
5. Steroid-dependent patients
6. Previous Tracheostomy

Exclusion criteria:

1. BMI<30
2. Thoracotomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1869 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartzell V Schaff, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Group | Retrospective Arm
Started | 272 | 1597
Completed | 272 | 1597
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Group | Retrospective Arm | Total
Number analyzed (Participants) | 272 | 1597 | 1869
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.4) | 65.7 (12.4) | 64.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 518 | 611
  Male | 179 | 1079 | 1258
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 272 | 1597 | 1869

OUTCOME MEASURES:

1. Primary Outcome: Wound Infection After Open Heart Surgery
Description: The total number of participants with surgical site infections after cardiac surgery.
Time Frame: 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Group | Retrospective Arm
Number analyzed (Participants) | 272 | 1597
Participants | 4 | 17
Statistical Analysis 1: Comparison: Prospective Group vs Retrospective Arm; Test type: Superiority; p = 0.55, Fisher Exact

2. Secondary Outcome: Reoperation for Wound Infection
Description: The total number of reoperations required due to infection.
Time Frame: 30 days post surgery
Population: Data on reoperation was not collected.
Arm/Group | Prospective Group | Retrospective Arm
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Length of Stay
Description: Length of stay was defined as the number of nights spent in the hospital after surgery.
Time Frame: postoperative to discharge
Population: Data for this outcome measure was not collected.
Arm/Group | Prospective Group | Retrospective Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 30 days postoperatively.
Arm/Group | Prospective Group | Retrospective Arm
All-Cause Mortality (participants affected / at risk) | 0/272 | 0/1597
Serious Adverse Events (participants affected / at risk) | 0/272 | 0/1597
Other Adverse Events (participants affected / at risk) | 0/272 | 0/1597

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02020018/Prot_SAP_000.pdf